CLINICAL TRIAL: NCT04107636
Title: Minimal Invasive Breast Cancer Excision Using Vacuum Assisted Biopsy Under Ultrasound Guidance
Acronym: MINIVAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); The Netherlands Cancer Institute (Other); St. Antonius Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL68820.091.19
Record Dates: First submitted 2019-06-13; First posted 2019-09-27 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Minimal invasive; Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assigned Interventions (Experimental): First, the tumor will be removed under local anesthesia using the VAB system with US guidance, through a small skin incision (<0.5 cm). A localization marker will be placed in the biopsy cavity, to help determine the cavity location. After 3 weeks, the breast conserving surgery is performed, excising the VAB excision cavity and a ≥1 cm of surrounding tissue, as deemed appropriate by the attending breast surgeon. A sentinel node biopsy will be performed in the same procedure.
  Interventions: Procedure: Vacuum assisted biopsy; Procedure: conventional lumpectomy

INTERVENTIONS:
Procedure: Vacuum assisted biopsy — First, the tumor will be removed under local anesthesia using the VAB system with US guidance, through a small skin incision (<0.5 cm). A localization marker will be placed in the biopsy cavity, to help determine the cavity location.
Procedure: conventional lumpectomy — After 3 weeks, the breast conserving surgery is performed, excising the VAB excision cavity and a ≥1 cm of surrounding tissue, as deemed appropriate by the attending breast surgeon. A sentinel node biopsy will be performed in the same procedure.

SUMMARY:
This study will assess whether it is feasible to remove small breast cancers completely using the Vacuum Assisted Biopsy (VAB) system System under Ultrasound guidance.

DETAILED DESCRIPTION:
Rationale: In the Netherlands, ≥7000 women undergo surgery for small breast cancers (T1) every year. In this study, the investigators will evaluate under which conditions it is possible to excise small breast cancers using the vacuum assisted biopsy (VAB) system under ultrasound (US) guidance. When successful, this can allow outpatient treatment of a selection of women with small breast cancers, improving the cosmetic outcome and quality of life.

Objective: Our study aim is to assess whether it is feasible to remove small breast cancers completely using the VAB system under US guidance.

Study design: This is a multi-centre, translational clinical phase II study in 170 women with cancers ≤15 mm based upon US and MRI measurements, and without mammographic or magnetic resonance imaging (MRI) evidence of more extensive disease (e.g. microcalcifications or non-mass enhancement).

Study population: Women with non-lobular invasive carcinomas, ≤15 mm based upon US and MRI measurements, no mammographic evidence of more extensive disease (e.g. microcalcifications or extensive architectural distortion), and sufficient space (roughly ≥6 mm, present or creatable by injection of saline) between the tumor and the dermis, nipple or pectoral muscle, are eligible for this study.

Intervention: In 170 women with cancers ≤15 mm based upon US and MRI measurements, and without mammographic evidence of more extensive disease (e.g. microcalcifications), after informed consent has been obtained, patients will be asked to fill out a questionnaire for assessment of breast cancer risk, using the Tyrer-Cuzick (or IBIS) model.

First, the tumor will be removed under local anesthesia using the VAB system with US guidance, through a small skin incision (<0.5 cm). A localization marker will be placed in the biopsy cavity, to help determine the cavity location. After 3 weeks, the breast conserving surgery is performed, excising the VAB excision cavity and a ≥1 cm of surrounding tissue, as deemed appropriate by the attending breast surgeon. A sentinel node biopsy will be performed in the same procedure.

Main study parameters/endpoints: Main endpoint of the study is the incidence of successful complete tumor excision by the VAB system, where successful is defined as having no tumor foci beyond 1 cm from the edge of the VAB cavity in the surgical re-excision specimen.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Our approach allows testing the feasibility of an innovating approach to remove breast cancer, with minimal negative effects or possible complications.

The burden from this study to the participating patients is the fact that two procedures are mandatory. This will result in prolonged time from initial diagnosis to end of surgical treatment. Positive study outcomes can pave the way to minimal invasive treatment in a selection of women, presenting with small breast tumors.

ELIGIBILITY:
Inclusion Criteria:

* Female sex.
* 18 years or older.
* US visible breast cancer.
* Histologically proven non-lobular invasive breast carcinoma with maximum diameter of 15 mm as assessed by US.
* Willing and able to undergo preoperative breast MRI
* Able to fill out the questionnaire
* Able to provide informed consent.

Exclusion Criteria:

* Male sex.
* 17 years or younger.
* No proven invasive breast cancer.
* Poor US visibility of the breast cancer.
* Neoadjuvant therapy.
* Contra-indications to breast MRI or intravenous contrast administration.
* Unable to fill out the questionnaire
* Unable to provide informed consent.
* Patients with breast implants.
* Pregnancy.
* Presence of additional malignant lesions at ipsilateral site on MRI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of successful complete tumor excision by the VAB system | Through study completion, an average of two months
  Successful is defined as 'having no residual (in situ) cancer in the surgical specimen'.

SECONDARY OUTCOMES:
Incidence of successful complete resection of the tumor based upon imaging related features using a questionnaire filled in by a radiologist. | 2 years
  An analysis will be performed to identify predicting factors for underestimation and for complete excision of the lesion after VAB. Factors included in the analysis are imaging related features from mammography, ultrasound and MRI (a.o. breast density, lesion type, shape, (background) enhancement). The questionnaire will be filled in by a radiologist.
Incidence of successful complete resection of the tumor based upon patient related features using a questionnaire filled in by the patient. | 2 years
  An analysis will be performed to identify predicting factors for underestimation and for complete excision of the lesion after VAB. Factors included in the analysis are patient related variables (a.o. age, body mass index, age at menarch, obstetric history, menopause status, history of a benign breast condition, history of ovarian cancer, use of hormone replacement therapy, family history). Patients will be asked to fill out a questionnaire for assessment of breast cancer risk, using the Tyrer-Cuzick (or IBIS) model.
Incidence of successful complete resection of the tumor based upon histopathological features from the large core biopsy specimens using a questionnaire filled in by a pathologist. | 2 years
  An analysis will be performed to identify predicting factors for underestimation and for complete excision of the lesion after VAB. Factors included in the analysis are histopathological related features from the large core biopsy specimen (a.o. type of cancer, vascular invasion, receptor status, grade). The questionnaire will be filled in by a pathologist.
Incidence of successful complete resection of the tumor based upon histopathological features from the VAB specimens using a questionnaire filled in by a pathologist. | 2 years
  An analysis will be performed to identify predicting factors for underestimation and for complete excision of the lesion after VAB. Factors included in the analysis are histopathological related features from the VAB specimen (a.o. type of cancer, vascular invasion, receptor status, grade, tubular formation, mitotic count). The questionnaire will be filled in by a pathologist.
Incidence of successful complete resection of the tumor based upon histopathological features from the surgical specimens using a questionnaire filled in by a pathologist. | 2 years
  An analysis will be performed to identify predicting factors for underestimation and for complete excision of the lesion after VAB. Factors included in the analysis are histopathological related features from the surgical specimen (a.o. type of cancer, vascular invasion, receptor status, grade, tubular formation, mitotic count, tumor satellites). The questionnaire will be filled in by a pathologist.
Analyze the difference in quality-of-life and pain experience between VAB excision and surgery. | 1 week
  In order to analyze the quality-of-life and differences in pain experience after VAE and surgery, patients will be asked to indicate a quality-of-life and pain experience score on the following time points:
  * 1 week after the VAB procedure.
  * 1 week following the surgical procedure.
  The EORTC QLQ-C30 questionnaire will be used to measure quality-of-life. All of the scales range from 1 to 4 or 1 to 7. A high scale score represents a higher response level. Thus a high score for the quality-of-life represents a high quality-of-life.

CONTACTS AND LOCATIONS:
Overall Officials: Ritse Mann, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands